CLINICAL TRIAL: NCT03444688
Title: Development and Evaluation of a Novel Portable Robotic Gait Rehabilitation Platform in Older Chronic Stroke Survivors (Phase 2)
Brief Title: Development and Evaluation of a Novel Portable Robotic Gait Rehabilitation in Chronic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSRB 2017/00696
Record Dates: First submitted 2018-01-28; First posted 2018-02-23 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-01

CONDITIONS: Stroke
Keywords: Robotic Walker
MeSH Terms: conditions — Stroke | interventions — Walkers

STUDY DESIGN:
Intervention Model Description: The recruited subjects will be divided into 2 groups through a simple randomization scheme using Microsoft Excel ("rand function"); 1) Conventional gait training (CT, control group) and 2) Gait rehabilitation with the new walker modified after 1st stage (WT, experimental group). Each subject will undergo training programs consisting of 45 minutes training session (excluding rest periods), 3 days (alternate) a week for 6 consecutive weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT, Control Group (Active Comparator): Conventional Gait Training
  Interventions: Other: Conventional Gait Training
- WT, Experimental Group (Experimental): Gait rehabilitation with walker
  Interventions: Device: Gait rehabilitation with walker

INTERVENTIONS:
Other: Conventional Gait Training — Subjects allocated to the CT group will first perform active assisted or passive range of motion of the lower limbs including ankle, knee, and hip joint in the supine position for 10 minutes. They will then perform conventional gait and balance therapy based on the proprioceptive neuromuscular facilitation (PNF) concept for 15 minutes. They will be given a 5 minutes rest. Finally, the CT subjects will undergo the over-ground gait training with or without aid or orthoses and with manual assistance from senior physiotherapist for 15 minutes, depending on the individual subject's abilities.
  Arms: CT, Control Group
Device: Gait rehabilitation with walker — For WT group, subjects will first go through active assisted or passive range of motion of the lower limbs including ankle, knee, and hip joint in the supine position for 10 minutes. The main therapy consists of 2 parts with 5 minutes rest in between. During part 1, subjects will be trained on the robotic walker with the help of active body weight support (BWS) and functional electrical stimulation (FES) for 15 minutes with pelvic motion support function and lateral balance function being continuously provided. During part 2, subjects will also receive resistance/assistance forces on top of the BWS and FES training for 15 minutes.
  Arms: WT, Experimental Group

SUMMARY:
The aims of this study is to test the training effects of the robotic walker. This study will compare the effectiveness of 2 different types of gait training protocols in chronic stroke patients, 1) conventional gait training (CT, control group), and 2) gait rehabilitation with the new walker modified after 1st stage (WT, experimental group).

DETAILED DESCRIPTION:
This will be a prospective single blind randomized control trial where investigators propose to recruit a maximum of 100 older chronic stroke patients (age 50 years to 90 years old) with mild to severe lower limb motor function impairment.

Recruited subjects will have 19 study visits. The recruited 100 subjects will be divided into 2 groups of 50 each through a simple randomization scheme; 1) Conventional gait training (CT, control group) and 2) Gait rehabilitation with the new walker modified after 1st stage (WT, experimental group). Each subject will undergo training programs consisting of 45 minutes training session (excluding rest periods), 3 days (alternate) a week for 6 consecutive weeks.

Subjects allocated to the CT group will receive physiotherapy program, including active assisted or passive range of motion and conventional gait and balance training. The subjects will first perform active assisted or passive range of motion of the lower limbs including ankle, knee, and hip joint in the supine position for 10 minutes. Subjects will then perform conventional gait and balance therapy based on the proprioceptive neuromuscular facilitation (PNF) concept for 15 minutes. Among the PNF techniques, investigators will facilitate pelvic motion to improve control and mobility of the subjects. Subjects will be given a 5 minutes rest. Finally, the CT subjects will undergo the over-ground gait training with or without aid or orthoses and with manual assistance from senior physiotherapist for 15 minutes, depending on the individual subject's abilities.

For WT group, subjects will first go through active assisted or passive range of motion of the lower limbs including ankle, knee, and hip joint in the supine position for 10 minutes. The main therapy consists of 2 parts with 5 minutes rest in between. During part 1, subjects will be trained on the robotic walker with the help of active body weight support (BWS) and functional electrical stimulation (FES) for 15 minutes with pelvic motion support function and lateral balance function being continuously provided. The level of BWS will be provided as much as the subjects can support his or her residual body weight (10% to 30% BWS). The BWS force will be gradually reduced as soon as the subjects can support his or her full body weight. The clinical criterion for the reduction is that the subjects show the ability to move his or her hips and are able to support his or her own body weight sufficiently on the affected lower limb and straighten their legs during the single-leg stance phase. Therapists will be able to control the level of BWS force according to the criteria mentioned above. FES will be used to stimulate the peroneal nerve in the affected side, and the intensity of the device will be painlessly controlled by allowing sufficient dorsiflexion and eversion during the swing phase. FES will be set to synchronize with the inertial measurement unit (IMU) sensors and the stimulation timing for the common peroneal nerve will based on the detected gait phase by IMU sensors. During part 2, subjects will also receive resistance/assistance forces on top of the BWS and FES training for 15 minutes. The decision on providing resistance or assistance modes will be made according to the subjects' functional ambulation category (FAC) level. For subjects with FAC level less than 3, the assistive function will be implemented, otherwise resistive function will be applied. The assistance and resistance forces will be applied proportional to the BW of the subjects (2% to 7% of BW), which is determined by therapists. The rationale of dividing the WT group into 2 parts of different training is that the 1st part is to provide basic locomotive function with persistent and repetitive sensory stimulation while the 2nd part is to add task-specificity to improve weight-bearing, aerobic, functional strengthening and balance for the neurologically challenged patients by implementing a variety of walking tasks. Investigators expect that the repetitive and persistent walking with task-specific gait training will promote better functional outcomes than the conventional gait therapy.

During the session, subjects can request for a rest anytime if they experience discomfort or fatigue. Additionally, investigators will provide them with a 5 - 15 minutes of rest time. The rest period given depends on individual subjects' needs. Investigators will seek their opinion whether subjects have enough rest and are well to continue with the session. Longer rest period will be given to the subjects who require them. During the resting period and also the period where subjects are not required to participate, a chair will be provided for the subject to sit and rest.

The session will be conducted under the supervision/assistance of senior physiotherapist, research assistants and engineering group. Clinical symptoms/adverse clinical developments will be closely monitored.

Outcomes will be measured before (T0), immediately after (T1) and 1 month after the end of treatment (T2) of 6 weeks therapy session by an independent senior physiotherapist to ensure blinding.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 50 years to 90 years old
* More than 6 months from first ever stroke but within 5 years confirmed by CT or MRI Brain
* Mild to severe unilateral motor weakness (hemiparesis has to be severe with lower extremity strength graded as 3 or less on the Medical Research Council scale in more than 2 muscle groups) and severity should be between 5 and 25 calculated according to National Institute of Health Stroke Scale
* Significant gait deficits ( Functional Ambulation Category , FAC ≤ 4 )
* Able to understand instructions and participate in rehabilitation
* Spasticity: Modified Ashworth Scale (MAS) less than 4
* Independent trunk control
* Comfortable to walk without a walking aid

Exclusion Criteria:

* Patient undergoing any formal rehabilitation program
* Multiple stroke
* Intracranial bleeds
* Any chronic disabling pathologies
* Spasticity limiting lower extremity ROM to less than 80 %
* Mini Mental State Examination (MMSE) score < 24
* Significant sensory deficit/ hemisensory neglect
* Any recent surgeries including orthopedic
* Active cancers or any other terminal illness
* Significant orthostatic hypotension
* Hip, knee and ankle arthrodesis
* Severe vascular disorders in lower limbs
* Having permanent pacemakers or ventriculoperitoneal shunt
* Subject's weight > 75kg

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-12-10 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | 3 minutes
  Modified Ashworth Scale (MAS) measures resistance during passive soft-tissue stretching. It is a quick and easy measure that can help assess the efficacy of treatment.
  MAS is performed in the supine position (this will garner the most accurate and the lowest score as any tension anywhere in the body will increase spasticity).
  Scoring 0 = Normal tone, no increase in tone 1 = Slight increase in muscle tone, manifested by a catch and release or minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion or extension
  1+ = Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 = More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved 3 = Considerable increase in muscle tone, passive movement difficult 4 = Affected part(s) rigid in flexion or extension
Medical Research Council (MRC) grading | 5 minutes
  The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
Functional Ambulation Category (FAC) | 2 minutes
  FAC is a functional walking test that evaluates ambulation ability.
National Institute of Health Stroke Scale (NIHSS) | 12 minutes
  NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Timed Up and Go (TUG) | 8 minutes
  TUG is a simple test used to assess a person's mobility and requires both static and dynamic balance.
Berg Balance Scale (BBS) | 15 minutes
  The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks. It is a valid instrument used for evaluation of the effectiveness of interventions and for quantitative descriptions of function in clinical practice and research.
  Description:
  14-item scale designed to measure balance of the older adult in a clinical setting.
  Equipment needed:
  Ruler, two standard chairs (one with arm rests, one without), footstool or step, stopwatch or wristwatch, 15 ft walkway
  Completion:
  Time: 15-20 minutes Scoring: A five-point scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56
  Interpretation:
  41-56 = low fall risk 21-40 = medium fall risk 0 -20 = high fall risk
  A change of 8 points is required to reveal a genuine change in function between 2 assessments.
Clinical Outcomes Variables Score (COVS) | 20 minutes
  The COVS assesses functional mobility across a broad range of neurologic conditions.
6 minute walk test | 6 minutes
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Temporal spatial gait analysis (Part 1) | 10 minutes
  Gait analysis is assessed by Tekscan Strideway which can provide temporospatial parameters including step length (cm), step width (cm), step time (s), step velocity (cm/s) and stride length (cm).
Temporal spatial gait analysis (Part 2) | 10 minutes
  Gait analysis is assessed by Tekscan Strideway which can provide temporospatial parameters including stride time (s), gait cycle time (s), stance time (s), swing time (s), single support time (s), and double support time (s).
Electromyography (EMG) | 10 minutes
  Electromyography (EMG) is evaluated by Delsys Trigno Wireless System which is a non-invasive method to detect muscle activity in mircoamperes. EMG sensors will be placed on Rectus Femoris, Tibilatis Anterior, Biceps Femoris, and lateral Gastrocnemius.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | 8 minutes
  Functional Independence Measure (FIM) is an 18-item of physical, psychological and social function. The tool is used to assess a patient's level of disability as well as change in patient status in response to rehabilitation or medical intervention.
  Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7.
  1. - Total assistance with helper
  2. - Maximal assistance with helper
  3. - Moderate assistance with helper
  4. - Minimal assistance with helper
  5. - Supervision or setup with helper
  6. - Modified independence with no helper
  7. - Complete independence with no helper
  Total score for the FIM motor subscale (the sum of the individual motor subscale items) will be a value between 13 and 91.
  Total score for the FIM cognition subscale (the sum of the individual cognition subscale items) will be a value between 5 and 35.
  Total score for the FIM instrument (the sum of the motor and cognition subscale scores) will be a value between 18 and 126.
Revised Nottingham Sensory Assessment (rNSA) | 15 minutes
  rNSA is a sensory assessment.
Number of falls | 1 year
  In the whole study, if there is more than 20% fall incidence, then the study will be compromised.
Patient's attitudes towards the robotic walker using visual analogue scale (EQ-5D VAS) ranging from 0 (negative) to 10 (positive). | 5 minutes
  EQ-5D VAS is a standardized instrument for measuring generic health status. The EQ-5D VAS essentially consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The subject is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.
  The EQ VAS records the subject's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the subject's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Santhosh Kumar Seetharaman, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt H, Sorowka D, Hesse S, Bernhardt R. [Development of a robotic walking simulator for gait rehabilitation]. Biomed Tech (Berl). 2003 Oct;48(10):281-6. doi: 10.1515/bmte.2003.48.10.281. German. PMID 14606269
- [Background] Patton J, Brown DA, Peshkin M, Santos-Munne JJ, Makhlin A, Lewis E, Colgate EJ, Schwandt D. KineAssist: design and development of a robotic overground gait and balance therapy device. Top Stroke Rehabil. 2008 Mar-Apr;15(2):131-9. doi: 10.1310/tsr1502-131. PMID 18430678
- [Background] Hornby TG, Campbell DD, Kahn JH, Demott T, Moore JL, Roth HR. Enhanced gait-related improvements after therapist- versus robotic-assisted locomotor training in subjects with chronic stroke: a randomized controlled study. Stroke. 2008 Jun;39(6):1786-92. doi: 10.1161/STROKEAHA.107.504779. Epub 2008 May 8. PMID 18467648
- [Background] Kwakkel G, Kollen BJ, Krebs HI. Effects of robot-assisted therapy on upper limb recovery after stroke: a systematic review. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):111-21. doi: 10.1177/1545968307305457. Epub 2007 Sep 17. PMID 17876068
- [Background] Mayo NE, Wood-Dauphinee S, Ahmed S, Gordon C, Higgins J, McEwen S, Salbach N. Disablement following stroke. Disabil Rehabil. 1999 May-Jun;21(5-6):258-68. doi: 10.1080/096382899297684. PMID 10381238
- [Background] Forster A, Young J. Incidence and consequences of falls due to stroke: a systematic inquiry. BMJ. 1995 Jul 8;311(6997):83-6. doi: 10.1136/bmj.311.6997.83. PMID 7613406
- [Background] Daly JJ, Zimbelman J, Roenigk KL, McCabe JP, Rogers JM, Butler K, Burdsall R, Holcomb JP, Marsolais EB, Ruff RL. Recovery of coordinated gait: randomized controlled stroke trial of functional electrical stimulation (FES) versus no FES, with weight-supported treadmill and over-ground training. Neurorehabil Neural Repair. 2011 Sep;25(7):588-96. doi: 10.1177/1545968311400092. Epub 2011 Apr 22. PMID 21515871
- [Background] Scheidt RA, Stoeckmann T. Reach adaptation and final position control amid environmental uncertainty after stroke. J Neurophysiol. 2007 Apr;97(4):2824-36. doi: 10.1152/jn.00870.2006. Epub 2007 Jan 31. PMID 17267755
- [Background] Patton JL, Stoykov ME, Kovic M, Mussa-Ivaldi FA. Evaluation of robotic training forces that either enhance or reduce error in chronic hemiparetic stroke survivors. Exp Brain Res. 2006 Jan;168(3):368-83. doi: 10.1007/s00221-005-0097-8. Epub 2005 Oct 26. PMID 16249912
- [Background] Kao PC, Srivastava S, Agrawal SK, Scholz JP. Effect of robotic performance-based error-augmentation versus error-reduction training on the gait of healthy individuals. Gait Posture. 2013 Jan;37(1):113-20. doi: 10.1016/j.gaitpost.2012.06.025. Epub 2012 Jul 24. PMID 22832470